CLINICAL TRIAL: NCT01444560
Title: The miRNA Machinery in Melanoma, Melanoma Metastases and Benign Melanocytic Naevi
Brief Title: miRNA Machinery in Melanoma, Melanoma Metastases and Benign Melanocytic Naevi
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Postdoc, Ruhr University of Bochum
Other Study IDs: microRNA4
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Cutaneous Melanoma; Nevi
MeSH Terms: conditions — Melanoma; Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — human skin
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Cutaneous Melanoma
- Cutaneous Melanoma Metastases
- Benign Melanocytic Nevi

SUMMARY:
MicroRNAs (miRNAs) are very small endogenous RNA molecules about 22-25 nucleotides in length, capable of post-transcriptional gene regulation. miRNAs bind to their target messenger RNAs (mRNAs), leading to cleavage or suppression of target mRNA translation based on the degree of complementarity. miRNAs have recently been shown to play pivotal roles in diverse developmental and cellular processes and linked to a variety of skin diseases and cancers. In the present study, the investigators examines the expression profiles of miRNA machinery components such as miRNA maturation and transport factors, microprocessor complex and RISC subunits in cutaneous melanoma, cutaneous melanoma metastases and benign melanocytic nevi.

DETAILED DESCRIPTION:
Patients with cutaneous melanoma, cutaneous melanoma metastases and benign melanocytic nevi were included in the study. Punch biopsies were harvested from the center of the tumors. The miRNA machinery components were detected by quantitative real-time reverse transcriptase polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* cutaneous melanoma
* cutaneous melanoma metastases
* benign melanocytic nevi

Exclusion Criteria:

* other forms of malignancy

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cutaneous melanoma, cutaneous melanoma metastases, benign melanocytic nevi
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2008-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Falk G Bechara, PD Dr., Study Director — Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum
Locations (1):
- Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Skrygan M, Georgas D, Sand D, Gambichler T, Altmeyer P, Bechara FG. The miRNA machinery in primary cutaneous malignant melanoma, cutaneous malignant melanoma metastases and benign melanocytic nevi. Cell Tissue Res. 2012 Oct;350(1):119-26. doi: 10.1007/s00441-012-1446-0. Epub 2012 Jun 17. PMID 22706980